CLINICAL TRIAL: NCT00181077
Title: Hypertonic Saline Use for Volume Expansion in Postpartum Preeclampsia
Brief Title: Hypertonic Saline Use in Preeclampsia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Abimbola Aina, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03--03-13-06
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Preeclampsia
Keywords: preeclampsia, hypertonic saline, diuresis
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 2% buffered hypertonic saline administration

SUMMARY:
To compare hypertonic saline to Lactated Ringer's solution and assess whether one speeds up the process of getting rid of extra body water faster in women with preeclampsia.

DETAILED DESCRIPTION:
Our patient population will consist of postpartum women who were diagnosed with preeclampsia in the antepartum period. Our goal is to enroll ten patients in the treated group and ten patients in the control group. The treatment group will have a 2% buffered hypertonic saline solution infused at 30 mL/hr in addition to receiving magnesium sulfate for seizure prophylaxis. The control group will receive the currently practiced regimen of infusion of a Lactated Ringer's solution at 75cc/hr. Both groups will be monitored on our Labor and Delivery unit as is the norm for any patient on a magnesium sulfate infusion. They will receive routine nursing care and hourly collaborative team assessments by the nurses and the physicians for signs of magnesium toxicity. Urine input/output ratios are evaluated on an hourly basis and a lung examination is performed to assess for pulmonary edema. A pulse oximeter will be used to obtain an hourly assessment of the patient's oxygenation status.

Both groups will have blood work evaluation every six hours for platelet count, electrolytes, liver enzymes, interleukin-1 and interleukin-6 (as markers of inflammation). We will collect information on patient symptoms regarding headache, visual changes and epigastric pain at 4-hour intervals and obtain the patient's weight immediately postpartum as well as at 24-hour intervals. Magnesium sulfate infusions will be discontinued at 24 hours postpartum or later at the discretion of the treating physician. No antihypertensive medications will be withheld from either group. Blood pressure will be obtained in the patients at the current interval of 60 minutes.

Hypertonic saline will be infused until the patient is 24 hours postpartum. Our primary outcome variable is the ratio of fluid intake to urine output. Data will be collected during the length of stay on our Labor and Delivery unit before the patient meets criteria for transfer to our postpartum unit, and their overall hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Women must have satisfied conditions for the diagnosis of preeclampsia (BP > 140/90, proteinuria ≥ 2+ or 300 mg in 24 hours)
* Women must have creatinine level below 1.6 mg/dL
* Women must have delivered their infant(s) prior to initiating therapy
* Women must be English-speaking
* Women must be medically stable at the time of entry into the study
* Women must be over the legal consenting age of 18 years
* Women must be consented prior to the administration of narcotics or other medications that may interfere with ability to give informed consent
* If not consented at the time of admission to Labor and Delivery, women must be comfortable enough with their contractions to complete the informed consent process without duress, or must be comfortable with regional anesthesia
* Women on magnesium sulfate will be eligible for entry after assessment of level of consciousness is deemed sufficient to give informed consent

Exclusion Criteria:

* Women not able to understand the study because of language barriers or significant learning impairment
* Women less than 18 years of age
* Women who are medically unstable prior to recruitment or in whom expeditious delivery is warranted
* Women who have developed eclampsia (or seizures as a result of their preeclamptic condition)
* Women who have not consented prior to the administration of narcotics or other medications that may interfere with their ability to give informed consent
* Women whose pain severity in labor is such that they cannot participate in informed consent
* Women with a pre-existing cardiomyopathy
* Women with a sodium level < 130, or > 150 mEq/L
* Women with a creatinine level greater than 1.6 mg/dL
* Women with co-morbid conditions that affect renal function i.e. lupus nephritis, diabetic nephropathy, or pre-existing hypertensive kidney disease
* Women whose level of consciousness on magnesium sulfate is deemed insufficient to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Fluid input to output ratios

SECONDARY OUTCOMES:
laboratory evaluation of inflammatory parameters (platelet count, IL-1, IL-6), liver enzymes, weight

CONTACTS AND LOCATIONS:
Overall Officials: Abimbola Aina-Mumuney, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland